CLINICAL TRIAL: NCT02302131
Title: Pulmonic SAPIEN XT™ THV A Multi-center, Observational Registry With Retrospective Enrollment of Patients That Underwent Transcatheter Pulmonic Valve Implantation and a Retrospective or Prospective Follow-up
Brief Title: Pulmonic SAPIEN XT THV
Acronym: Pulmonic XT
Status: Completed | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Estimate, GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: EU Pulmonic XT
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Valve Malfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pulmonary valve replacement: SAPIEN XT Transcatheter Heart Valve in the pulmonic position at the time of data collection
  Interventions: Other: SAPIEN XT

INTERVENTIONS:
Other: SAPIEN XT — Patients that have undergone percutaneous implantation of an Edwards SAPIEN XT Transcatheter Heart Valve in the pulmonic position at the time of data collection

SUMMARY:
Multi-center, Observational Registry with Retrospective Enrollment and Prospective Follow-up.

The aim of the registry is to document the feasibility and safety of implanting an Edwards SAPIEN XT transcatheter heart valve in the pulmonic position.

DETAILED DESCRIPTION:
A malfunction or dysplasia of the pulmonary valve or the right ventricular outflow tract (RVOT) is one of the major components of the cardiac physiology in many congenital heart defects. Surgical correction of complex heart defects often includes some form of surgical repair or replacement of the native RVOT by biological valves such as homograft, bioprosthesis or Xenografts (i.e., Contegra conduits). Typical examples are tetralogy of Fallot (TOF) or double outlet right ventricle (DORV), pulmonary stenosis (PS), pulmonary atresia (PA), truncus arteriosus (TA), transposition of the great arteries (TGA) with PS (Rastelli's operation), absent pulmonary valve syndrome (Miller-Lev-Paul), Ross surgery for aortic valve disease and others. The repaired or replaced pulmonary valve however often becomes dysfunctional later on and many patients require surgical revisions of the RVOT with pulmonary valve replacement within 10 years of primary intervention.

TPVI provides a less invasive alternative to surgery in patients with right ventricular-to-pulmonary artery (RV-PA) conduit dysfunction. Early results of percutaneous pulmonary valve implantation (PPVI) showed that it is a promising procedure compared to a conventional surgical intervention. Meanwhile, pre-stenting of the RVOT before PPVI is routinely performed, enabling PPVI in various anatomies.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication and decision for the implantation of an Edwards SAPIEN XT THV made
* Data release form

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have undergone percutaneous implantation of an Edwards SAPIEN XT Transcatheter Heart Valve in the pulmonic position at the time of data collection
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
right ventricular and pulmonary artery pressure | 30 days
max flow velocity RVOT | 30 days
NYHA class | 30 days
degree of pulmonary regurgitation | 30 days
procedural success | 30 days
Peak gradient | 30 days
length of hospitalization | 30 days
Peak Oxygen consumption | 24 months
anaerobic threshold | 24 months
device function | 24 months
structural valve Deterioration including stent fracture | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Haas, MD, Principal Investigator — Center for Congenital Heart Defects, Heart and Diabetes Center NRW; Peter Bramlage, MD, Principal Investigator — IPPMed
Locations (6):
- Belgium (2):
  - Gent University Hospital, Ghent
  - UZ Leuven, Leuven
- Canada (3):
  - St Pauls Hospital, Vancouver, British Columbia
  - Toronto General, Toronto, Ontario
  - Hospital Laval, Ste Foy, Montreal, Quebec
- Universitätshospital Zürich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Haas NA, Carere RG, Kretschmar O, Horlick E, Rodes-Cabau J, de Wolf D, Gewillig M, Mullen M, Lehner A, Deutsch C, Bramlage P, Ewert P. Early outcomes of percutaneous pulmonary valve implantation using the Edwards SAPIEN XT transcatheter heart valve system. Int J Cardiol. 2018 Jan 1;250:86-91. doi: 10.1016/j.ijcard.2017.10.015. Epub 2017 Oct 6. PMID 29017776